## **Randomized Controlled Study Protocol:**

Effect of Laughter Yoga on Mental Symptoms Frequency and Level of Saliva Cortisol

14/01/2019

Fatma Ozlem OZTURK\_RN, Ph. D., Ankara University Faculty of Nursing

Department of Nursing Altindag, Ankara-Turkey

Ayfer TEZEL RN, Ph.D. Professor Ankara University Faculty of Nursing

Department of Nursing Altindag, Ankara-Turkey

None conflict of interest statement

Please address all correspondence in regard to this article to: F. Ozlem Ozturk, Ph. D., Academician, Ankara University, Faculty of Nursing, Department of Nursing, Altindag, Ankara-Turkey.

E-mail: foozturk@ankara.edu.tr / fozlemozturk@gmail.com

Tel: +90-3123191450-1125

## **ANALYSİS**

Data analysis will be done in SPSS for Windows 14 package program. Number, percentage, mean, standard deviation, minimum and maximum values will be used as descriptive statistics. Data obtained in the groups will be given as mean  $\pm$  standard deviation. The chi-square test will be used to evaluate the differences in terms of sociodemographic characteristics, and the difference between the two means will be used in the evaluation of the difference between the two independent groups. The level of statistical significance will be accepted as p <0.05.